CLINICAL TRIAL: NCT02032082
Title: Rule of Carbone Monoxyde in the Ex Vivo Lung Perfusion Reconditionning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Asmae Belhaj, MD, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: EVLP-CO
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Neurogenic Lung Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Ex vivo without CO (No Intervention)
- EX Vivo with carbone monoxide (Experimental): During the Ex Vivo Lung Perfusion reconditioning,the lungs will be ventilated wit h Oxygen (21%) and Carbon Monoxide (250ppm).
  Interventions: Other: Carbone monoxide

INTERVENTIONS:
Other: Carbone monoxide
  Arms: EX Vivo with carbone monoxide

SUMMARY:
Ex vivo lung perfusion (EVLP) is not a new concept and has been widely used to study lung function in small animals. It also has been shown to be a useful technique to evaluate lungs from donation after cardiac death (DCD) (Yeung, Thorac Surg Clin, 2009). It has been recently demonstrated successful application of an acellular EVLP technique in optimalizing lung function ex vivo for an extended period of time. Following 12 h of normothermic EVLP, patients were transplanted and demonstrated immediate life-sustaining function with promising short-term evolution (Aigner, Am J Transplant, 2012; Sanchez, J Heart Lung Transplant, 2012; Cypel, N Engl J Med, 2011).

Lung donation obtained after carbon monoxide intoxication has been recognized as excellent organs because of less general inflammation and less primary graft dysfunction after procedure. In a murine model of brain dead, carbon monoxide inhalation at a low concentration (50 to 500 parts per million (ppm)) exerts significant cytoprotection in several lung injury models via its vasodilatation, anti-inflammatory, and anti-apoptotic properties (Dong, J Heart Lung transplant, 2010). The carbon monoxide inhalation down-regulates pro-inflammatory cytokines (TNF-alpha, IL-6) along with the increase of anti-inflammatory cytokine (IL-10) in recipient serum. The inhalation significantly decreases cell apoptosis in lung grafts, inhibiting mRNA and protein expression of intercellular adhesion molecule-1 (ICAM-1) and caspase-3 in lung grafts (Zhou, Chin Med J, 2008).

Apoptotis and inflammatory processes may, in part, concern alveolar tissue. Research in the field of biomarkers is now opening new perspectives with the development of non-invasive tests allowing for monitoring inflammation and damage in the deep lung. Blood tests (Bernard, Toxicol Appl Pharmacol, 2005) measuring lung-specific proteins (pneumoproteins) such as Clara cell protein (CC16) and surfactant-associated proteins (A, B or D) are now available to evaluate the permeability and/or the cellular integrity of the pulmonary epithelium. These dosages may constitute an interesting way for monitoring the quality of the lung before implantation.

ELIGIBILITY:
Inclusion Criteria:

Lung Edema

Exclusion Criteria:

Infection Severe Emphysema Tumor

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Incidence on Primary Graft Dysfunction | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Mont-Godinne, Yvoir, Namur, Belgium